CLINICAL TRIAL: NCT00044278
Title: An Open-Label, Uncontrolled, Long-Term Study to Assess the Safety of LAMICTAL in Pediatric Subjects Previously Enrolled in Protocol LAM20006 and In LAMICTAL-naive Subjects (1-24 Months of Age)
Brief Title: Pediatric Epilepsy Study in Subjects 1-24 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAM20007
Record Dates: First submitted 2002-08-23; First posted 2002-08-26 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Epilepsy
Keywords: epilepsy; pediatric; partial seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lamotrigine

SUMMARY:
This study will evaluate the long-term safety of LAMICTAL(lamotrigine)in subjects with partial seizures previously enrolled in protocol LAM20006 and in subjects 1-24 months of age who have never received LAMICTAL(LAMICTAL-naive). For LAMICTAL-naive subjects, LAMICTAL will be added to the subject's current epilepsy medications.

ELIGIBILITY:
Inclusion criteria:

* Must have completed the Open-Label Phase of protocol LAM20006 or meet criteria for LAMICTAL naive subjects as follows:
* A confident diagnosis of epilepsy.
* 4 or more partial seizures per month.
* current treatment with 1 or 2 anti-epileptic drugs.

Exclusion criteria:

* Has seizures not related to epilepsy.
* Has a surgically implanted and functioning vagal nerve stimulator.
* Has previously been treated with lamotrigine.
* Is currently taking felbamate, ACTH (adrenocorticotrophic hormone) or is on the ketogenic diet.
* Use of experimental medication within 30 days of enrollment.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 197 (Actual)
Dates: Start 2000-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with overall, serious, drug-related treatment emergent adverse events and adverse events leading to premature study discontinuation | 43 Months
Change from baseline in vital signs -heart rate (HR) | Up to 43 Months
Change from baseline in vital signs - weight (WT) | Up to 43 months
Change from baseline in vital signs - height (HT) | Up to 43 months
Change from baseline in vital signs - head circumference (HC) | Up to 43 months
Change from baseline in clinical chemistry parameters including Albumin and Total protein | Up to month 43
Change from baseline in clinical chemistry parameters including alkaline phosphatase, Alanine transaminase (ALT), and Aspartate Aminotransferase (AST) | Up to 43 moths
Change from baseline in clinical chemistry parameters including total bilirubin and creatinine | Up to 43 months
Change from baseline in clinical chemistry parameters including glucose (glu), potassium (K), sodium (Na) and urea | Up to 43 months
Change from baseline in hematological parameters including bands, basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and total white blood cells (WBC) | Up to 43 moths
Change from baseline in Hemoglobin (Hb) | Up to 43 months
Change from baseline in Mean corpuscular hemoglobin (MCH) | Up to 43 months
Change from baseline in Mean corpuscular hemoglobin concentration (MCHC) | Up to 43 months
Change from baseline in mean corpuscular volume (MCv) | Up to 43 months
Change from baseline in red blood cells (RBC) | Up to 43 months
Number of participants with treatment emergent neurological abnormalities | Up to 43 months
Number of participants with treatment emergent clinically significant ECG abnormalities | Up to 43 months
Number of participants with potentially clinically significant change in hematology parameters | Up to 43 months
Number of participants with potentially clinically significant change in clinical chemistry parameters | Up to 43 months
Number of participants with potentially clinically significant change in vital signs | Up to 43 months

SECONDARY OUTCOMES:
Mean percentage change in seizure frequency between the Historical Baseline Phase and over the course of the 48-week Treatment Phase | Up to 48 Weeks
Investigator's assessment of the participant's overall clinical status | Up to 43 months
Mean Maximal plasma concentration (Cmax) in serum and saliva of Lamicital -naïve participants | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (68):
- United States (39):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Morristown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Argentina (2):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- GSK Investigational Site, Parkville, Melbourne, Victoria, Australia
- GSK Investigational Site, Tartu, Estonia
- GSK Investigational Site, Reims, France
- Hungary (5):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Szeged
- Italy (6):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Mantova, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Messina, Sicily
  - GSK Investigational Site, Padua, Veneto
- GSK Investigational Site, Riga, Latvia
- GSK Investigational Site, Beirut, Lebanon
- GSK Investigational Site, Kaunas, Lithuania
- Netherlands (3):
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Portugal (3):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- GSK Investigational Site, SanJuan, Puerto Rico, Puerto Rico
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Prešov
- GSK Investigational Site, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: LAM20007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LAM20007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LAM20007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LAM20007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LAM20007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LAM20007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LAM20007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register